CLINICAL TRIAL: NCT03966456
Title: Real World Study of Immunotherapy-Comparison of Four PD-1 Agents in China
Brief Title: Real World Study of Four PD-1 Agents in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, zhangxiaochun, Director of Cancer Precision Medical Center, The Affiliated Hospital of Qingdao University
Other Study IDs: Ic-01
Record Dates: First submitted 2019-05-22; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Thoracic Cancer; Gynecologic Cancer; Abdomen Tumors; Malignant Melanoma
MeSH Terms: conditions — Abdominal Neoplasms; Melanoma | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- nivolumab: Consecutive patients treated with nivolumab single or combined chemotherapy/targeting therapy.
  Interventions: Drug: Chemotherapy
- pembrolizumab: Consecutive patients treated with pembrolizumab single or combined chemotherapy/targeting therapy.
  Interventions: Drug: Chemotherapy
- toripalimab: Consecutive patients treated with toripalimab single or combined chemotherapy/targeting therapy.
  Interventions: Drug: Chemotherapy
- sintilimab: Consecutive patients treated with sintilimab single or combined chemotherapy/targeting therapy.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — compare the effecy and safety of 4 PD-1 agents single and combined with chemotherapy in chinese people.
  Other Names: targeting therapy

SUMMARY:
Consecutive patients treated with PD-1 therapy in Qingdao City were included in our study. The effecy and safety of the four PD-1 agents according to clinical outcomes in real world will be studied.

DETAILED DESCRIPTION:
Consecutive patients treated with PD-1 therapy in Qingdao City were included in our study. The effecy and safety of the four PD-1 agents according to clinical outcomes in real world will be studied. ORR will be studied of the four PD-1 agents（nivolumab, pembrolizumab, toripalimab, sintilimab）

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung cancer, liver cancer and other solid cancers
* Histologically or cytologically confirmed diagnosis cancer treated with PD-1 agents
* At least one measurable lesion
* Eastern Cooperative Oncology Group (ECOG) Performance Scale 0 or 1 Adequate organ function

Exclusion Criteria:

* patients treated with PD-1 agents less than 2 terms

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients treated with PD-1 agents (nivolumab, pebrolizumab, toripalimab, sintilimab)
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 1 year
  ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters). The percentage of strongly PD-L1 positive participants who experienced a CR or PR is presented.

SECONDARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | 1 year
  Adverse events are defined as any adverse medical events that occur in the participants taking the drugs and do not necessarily have a causal relationship with the treatment.

OTHER OUTCOMES:
PFS | 2 years
  PFS was defined as the time from the first day of study treatment to the first documented disease progression per irRC or death due to any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Zhang, Dr, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
IPD only shared in the study group